CLINICAL TRIAL: NCT03725501
Title: A Phase 2, Multicenter, Randomized, Placebo-Controlled, Double-Blind, Three-arm Parallel-Group, 12-Month Study to Evaluate the Safety and Efficacy of ALS-L1023 Administered in Combination With Ranibizumab in Patients With Wet-AMD
Brief Title: Evaluation of the Safety and Efficacy of ALS-L1023 Administered in Combination With Ranibizumab in Patients With Wet-AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AngioLab, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALS-L1023_AMD_201
Record Dates: First submitted 2018-10-02; First posted 2018-10-31 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — ALS-L1023; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ranibizumab + ALS-L1023 600mg (Experimental): * ALS-L1023 600 mg - Take 2 tablets orally twice a day.
  * Ranibizumab (Lucentis®)
    * Loading Phase (3 months): Intravitreally inject 0.5 mg of Ranibizumab/0.05 mL monthly.
    * PRN Phase (9 months): It should only be administered to subjects who meet the re-administered criteria.
  Interventions: Drug: ALS-L1023; Drug: Ranibizumab
- Ranibizumab + ALS-L1023 1200mg (Experimental): * ALS-L1023 1200 mg - Take 2 tablets orally twice a day.
  * Ranibizumab (Lucentis®)
    * Loading Phase (3 months): Intravitreally inject 0.5 mg of Ranibizumab/0.05 mL monthly.
    * PRN Phase (9 months): It should only be administered to subjects who meet the re-administered criteria.
  Interventions: Drug: ALS-L1023; Drug: Ranibizumab
- Ranibizumab + Placebo (Placebo Comparator): * Placebo - Take 2 tablets orally twice a day.
  * Ranibizumab (Lucentis®)
    * Loading Phase (3 months): Intravitreally inject 0.5 mg of Ranibizumab/0.05 mL monthly.
    * PRN Phase (9 months): It should only be administered to subjects who meet the re-administered criteria.
  Interventions: Drug: Ranibizumab; Other: Placebo

INTERVENTIONS:
Drug: ALS-L1023 — ALS-L1023 is an active fraction extracted from Melissa officinalis L. (Labiatae; lemon balm) leaves.
  Other Names: McEye
  Arms: Ranibizumab + ALS-L1023 1200mg; Ranibizumab + ALS-L1023 600mg
Drug: Ranibizumab — LUCENTIS® (an anti-neovascular VEGF-A inhibitor) 0.5 mg, intravitreal injection
  Other Names: Lucentis
Other: Placebo — Control group for comparison with oral administration of ALS-L1023
  Arms: Ranibizumab + Placebo

SUMMARY:
The objective of this phase 2 study is to determine the optimal dose of ALS-L1023 by evaluating the safety and efficacy of ALS-L1023 comparing with placebo when used in combination with Ranibizumab for the treatment of wet age-related macular degeneration(AMD).

The study is designed as multicenter, randomized, placebo-controlled, double-blind, three-arm parallel-group phase 2 study in patients with neovascular age-related macular degeneration.

This study consists of two separate phases: a loading phase and a PRN(pro re nata) phase.

Once the subject provides a written informed consent, subject information including demographics, medical history, and concomitant medications will be collected, and only those who meet the inclusion/exclusion criteria will participate in the study.

All subjects who are enrolled in the study will be randomized into three groups Group A (Ranibizumab 0.5mg & ALS-L1023 600mg) or Group B (Ranibizumab 0.5mg & ALS-L1023 1200mg) or Group C (Ranibizumab & placebo) in a 1:1:1 ratio. Randomization will be stratified by whether or not the subject has PCV(polypoidal choroidal vasculopathy) confirmed at Screening test.

During the 3-month loading phase, all subjects will receive a Ranibizumab 0.5mg injection into the vitreous every month and take either the placebo or ALS-L1023 orally twice a day. During the following 3-12 month PRN phase, subjects will continue to take the placebo or ALS-L1023 in the same frequency as above but receive Ranibizumab injection only when it meets retreatment criteria. Subjects must instill antibacterial eye drops three times a day for three days after Ranibizumab injection.

Subjects will visit the study site monthly during the 12 month study period in order to receive scheduled assessments and evaluate safety and efficacy of treatment. Image interpretation will be performed by a central reading center. The central reading center will confirm eligibility for enrollment and the discrimination of Polypoidal Choroidal Vasculopathy(PCV) at screening and play a role in interpreting whole images of all subjects after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 50 years or older;
2. Subjects who can give a written informed consent;
3. Subjects who have active, subfoveal choroidal neovascularization(CNV) Active indicates the confirmation of fluorescence leakage by FAG and the presence of intraretinal or subretinal fluid by optical coherence tomography(OCT);
4. Subjects whose area of fibrosis is less than 50% of total lesion area;
5. Subjects with BCVA letter score of 73-24 (20/40 to 20/320 Snellen Equivalent) using ETDRS chart measured at 4 meters distance;
6. Subjects who have a maximum lesion size of 12 optic-disk areas (1 optic-disk area equals 2.54 mm2 on the basis of 1 optic-disk diameter of 1.8 mm) with neovascularization.

Exclusion criteria:

1. Subjects who have any prior ocular or systematic treatment or surgery in the study eye for neovascular AMD like Photodynamic therapy(PDT), laser photocoagulation etc. except dietary supplements or vitamins;
2. Subjects who received any prior or concomitant therapy in the study eye with anti-VEGF therapy (for example Ranibizumab, Bevacizumab, Aflibercept etc.). This does not apply to treatment of the opposite eye;
3. Subjects whose total lesion size is ≥12 disc areas (30.5 mm2), including blood, scars, and neovascularization) as assessed by Fluorescein angiography(FAG) in the study eye;
4. Subjects who have sub-retinal hemorrhage that is either 50% or more of the total lesion area, or if the blood is under the fovea and is 1 or more disc areas in size in the study eye (if the blood is under the fovea, then the fovea must be surrounded 270° by visible CNV);
5. Subjects who have scar or fibrosis making up >50% of the total lesion in the study eye;
6. Subjects who have scar, fibrosis, or atrophy involving the center of the fovea in the study eye;
7. Subjects who have presence of retinal pigment epithelial tears or rips involving the macula in the study eye;
8. Subjects with a history of any vitreous hemorrhage within 4 weeks prior to Screening in the study eye;
9. Subjects who have presence of other causes of CNV in the study eye;
10. Subjects who had prior vitrectomy in the study eye;
11. Subjects with a history of retinal detachment or treatment or surgery for retinal detachment in the study eye;
12. Subjects with any history of macular hole of stage 2 and above in the study eye;
13. Subjects who have any intraocular or periocular surgery within 3 months of Day 1 on the study eye, except lid surgery, which may not have taken place within 1 month of Day 1, as long as it is unlikely to interfere with the injection;
14. Subjects diagnosed with diabetes who have diabetic retinopathy or HbA1c value of 8 or more at screening;
15. Subjects with a history or clinical evidence of diabetic retinopathy, diabetic macular edema or any retinal vascular disease other than AMD in either eye;
16. Subjects who have macular disease or media opacity (including cataracts and vitreous opacity) that can be affect vision at the time of AMD diagnosis according to investigator' discretion;
17. Subjects who have hypersensitivity to investigational products or to drugs with similar chemical structures;
18. Subjects with infections/suspected infections in or around the eye;
19. Subjects who have severe intraocular inflammation;
20. Female subjects who are pregnant or breastfeeding;
21. Female subjects of childbearing age but are not using one or more of the following contraceptive methods:

    * Surgically sterile (i.e. have had bilateral tubal ligation or vasectomy)
    * Hormonal contraceptives (implant, patch, or oral)
    * Double barrier contraception (must use two of the following: intrauterine device, male or female condoms with spermicide, diaphragm, contraceptive sponge, cervical cap)
    * Periodic abstinence (i.e. calendar rhythm method, Billings Ovulation Method, and basal body temperature) and withdrawal method are not considered as appropriate contraceptive methods, and subjects must continue to use effective methods of contraception throughout the study and for 30 days after the end of the study;
22. Subjects who experienced cardiovascular or cerebrovascular events within 12 months prior to Screening;
23. Subjects who have any clinically significant medical condition that would interfere with the study outcomes or subjects who are deemed inappropriate to participate in the study according to Investigator's discretion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Mean change of Best Corrected Visual Acuity(BCVA). | 12 months
  Mean change of BCVA(Best Corrected Visual Acuity) as assessed by ETDRS(Early Treatment Diabetic Retinopathy Study) chart at a distance of 4 meters at month 12 compared with baseline.

SECONDARY OUTCOMES:
Mean change in BCVA(at each visit) | 12 months
  Mean change in BCVA as assessed by ETDRS chart at a distance of 4 meters at each visit except month 12 compared with baseline.
Mean number of Ranibizumab re-administration | 12 months
  Mean number of Ranibizumab re-administration after Ranibizumab loading dose.

CONTACTS AND LOCATIONS:
Overall Officials: SeWoong Kang, Study Chair — Samsung Medical Center
Locations (1):
- AngioLab, Inc., Daejeon, Daejeon Gwangyeogsi, South Korea

IPD SHARING:
Plan to Share IPD: No